CLINICAL TRIAL: NCT05346679
Title: DIABETES EATING PROBLEM SURVEY- REVISED (DEPS-R) AMONG ADULTS WITH TYPE 1 DIABETES
Brief Title: DEPS-R Turkish Version in Adults With Type 1Diabetes
Acronym: DEPS-R
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasemin Atik Altinok, Dietician, PhD, Ege University
Other Study IDs: DEPS-R Adult
Record Dates: First submitted 2022-04-16; First posted 2022-04-26 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; DEPS-R; confirmatory factor analysis; diabulimia; distributed eating disorder
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabulimia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A growing body of research has revealed the good psychometric properties and three-component factor structure of DEPS-R in children and adolescents with type 1 diabetes (T1D) but research with adults has limited and has differing results. The Diabetes Eating Problem Survey-Revised (DEPS-R) developed by Markowitz et al is a diabetes-specific self-report instrument to screen eating disorders for individuals with T1D. DEPS-R is a 16-item diabetes-specific self-report questionnaire to test for diabetes-specific eating disorders. Answers are scored on a six-point Likert scale, with higher scores indicating more DEB and a total score of ≥20 indicating a high risk for eating disorders (range 0-80). The original DEPS-R has been shown to have a good internal consistency (Cronbach's alpha=0.86) and construct validity in a sample of the pediatric population with T1D. This study aimed to evaluate the validity and reliability of the Turkish version of the DEPS-R questionnaire for adults with T1D, investigate its psychometric properties and factor structure, and examine its relationship with the EDE-Q questionnaire.

DETAILED DESCRIPTION:
In this cross-sectional study, participants answered a DEPS-R and EDE-Q questionnaire during a regularly scheduled medical visit after obtaining written informed consent. All participants had established that patients with T1D were treated with multiple daily insulin or insulin pump therapy. Height was measured using a stadiometer to the nearest 0.1 cm in all participants. Weight was measured unclothed to the nearest 0.1 kg using a calibrated balance scale. Body Mass Index (BMI) was calculated by using the weight (kg)/height (m²) equation. Clinical data including HbA1c, T1D onset, birth date, and treatment model etc. was conducted as part of a standard clinical assessment. HbA1c was measured with ion-exchange high-performance liquid chromatography (Bio-rad Variant ll Turbo, Japan).

ELIGIBILITY:
Inclusion Criteria:

* Duration of T1D ≥1 year
* A regular follow-up for at least 1 year (4 visits/year)
* No major medical problems related to nutrition

Exclusion Criteria:

* Have major medical problems related to nutrition ( etc. celiac disorders, cystic fibrosis, dyslipidemia,.....)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The sample of this study consists of 100 participants with T1D who were being followed at the Istanbul University, Istanbul Faculty of Medicine, Endocrine and Diabetes Outpatient Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
DEPS-R Score | Day 1
  Diabetes Eating Problem Survey-Revised, min score 0, max score 80 DEPS-R score DEP-R score ≥20 indicating a high risk for eating disorders
EDE-Q Score | Day 1
  Eating Disorders Examination Questionnaire It consists of four subscales eating restraint, eating concern, shape concern, and weight concern. The global score represents an average of the four subscale scores, with higher scores indicating greater eating pathology.
Duration of diabetes (years) | Day 1
  It will be calculated by subtracting the diabetes onset date from the date the patient was included in the study.
HbA1c | Day 1
  number
BMI | Day 1
  number

CONTACTS AND LOCATIONS:
Overall Officials: yasemin A atik-altınok, PhD, Study Chair — ege university department of pediatrics
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Atik Altinok Y, Ozgur S, Meseri R, Ozen S, Darcan S, Goksen D. Reliability and Validity of the Diabetes Eating Problem Survey in Turkish Children and Adolescents with Type 1 Diabetes Mellitus. J Clin Res Pediatr Endocrinol. 2017 Dec 15;9(4):323-328. doi: 10.4274/jcrpe.4219. Epub 2017 Feb 23. PMID 28270369
- [Background] Karastogiannidou C, Giannoulaki P, Samaras I, Kotzakioulafi E, Didangelos T, Bocsan IC, Vassilopoulou E. The Diabetes Eating Problem Survey-Revised (DEPS-R) in a Greek Adult Population with Type 1 Diabetes Mellitus: Model Comparison Supporting a Single Factor Structure. Nutrients. 2021 Jul 12;13(7):2375. doi: 10.3390/nu13072375. PMID 34371885
- [Background] Wisting L, Wonderlich J, Skrivarhaug T, Dahl-Jorgensen K, Ro O. Psychometric properties and factor structure of the diabetes eating problem survey - revised (DEPS-R) among adult males and females with type 1 diabetes. J Eat Disord. 2019 Jan 17;7:2. doi: 10.1186/s40337-018-0232-0. eCollection 2019. PMID 30675355
- [Background] Wisting L, Froisland DH, Skrivarhaug T, Dahl-Jorgensen K, Ro O. Psychometric properties, norms, and factor structure of the diabetes eating problem survey-revised in a large sample of children and adolescents with type 1 diabetes. Diabetes Care. 2013 Aug;36(8):2198-202. doi: 10.2337/dc12-2282. Epub 2013 Mar 27. PMID 23536586
- [Background] Yilmaz Kafali H, Atik Altinok Y, Ozbaran B, Ozen S, Kose S, Tahillioglu A, Darcan S, Goksen D. Exploring emotional dysregulation characteristics and comorbid psychiatric disorders in type 1 diabetic children with disordered eating behavior risk. J Psychosom Res. 2020 Apr;131:109960. doi: 10.1016/j.jpsychores.2020.109960. Epub 2020 Feb 11. PMID 32070835
- [Background] Watt A, Ng AH, Sandison A, Fourlanos S, Bramley A. Prevalence of disordered eating in adults with type 1 diabetes in an Australian metropolitan hospital. Health Soc Care Community. 2022 Jul;30(4):e974-e980. doi: 10.1111/hsc.13500. Epub 2021 Jul 12. PMID 34250682
- [Derived] Atik-Altinok Y, Eliuz-Tipici B, Idiz C, Ozgur S, Ok AM, Karsidag K. Psychometric properties and factor structure of the diabetes eating problem survey- revised (DEPS-R) among adults with type 1 diabetes mellitus. Eat Weight Disord. 2023 Sep 4;28(1):71. doi: 10.1007/s40519-023-01602-y. PMID 37665472